CLINICAL TRIAL: NCT00409565
Title: A Phase II Trial of Cetuximab and Bevacizumab in Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00171; NCI / CTEP Protocol # 7440; NCT00407810 (obsolete NCT alias)
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
Keywords: head and neck cancer; cetuximab; bevacizumab; squamous cell carcinoma; SCCHN; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab plus bevacizumab (Experimental): Cetuximab plus bevacizumab
  Interventions: Drug: Cetuximab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Cetuximab — * Cetuximab 400 mg/m2 IV over 120 minutes on day 1 of cycle 1 ONLY
  * Cetuximab dose will be 250 mg/m2 IV over 60 minutes weekly on ALL subsequent administrations
  Other Names: Erbitux, C225
Drug: Bevacizumab — Once every 3 weeks, 15 mg/kg of bevacizumab will be given by IV infusion after cetuximab has been given
  Other Names: (rhuMAb VEGF, Avastin) (NSC 704865; IND 7921)

SUMMARY:
The purpose of this study is to determine if the combination of two new drugs, cetuximab (Erbitux) and bevacizumab (Avastin) can increase the effectiveness of treatment for head and neck cancer. Cetuximab has recently been approved by the FDA for head and neck cancer (that is locally or regionally advanced) when used in combination with radiation therapy. Cetuximab is also approved by the FDA for the treatment of colorectal cancer

DETAILED DESCRIPTION:
Approximately 40,000 new cases of head and neck cancer are diagnosed annually in the United States 1. Squamous cell carcinomas account for more than 90% of head and neck cancer cases. Patients with squamous cell carcinoma of the head and neck (HNSCC) usually present with locoregionally advanced disease. Initial presentation with distant metastasis may occur in about 10% of all patients. However, recurrence of disease either in local or distant sites after potentially curative treatment with surgery, radiation, and/or chemotherapy occurs in more than 50% of patients. Therefore, the majority of patients with HNSCC develop recurrent or metastatic disease during the course of their illness. These patients have a dismal prognosis with a median survival of 6-9 months 2-4.

Active single agents in head and neck squamous cell carcinoma include methotrexate, bleomycin, cisplatin, carboplatin, 5-FU, paclitaxel, docetaxel, and CPT-11. A small randomized study showed that cisplatin monotherapy prolongs survival compared with best supportive care 5. Response rates for single agents range between 10-40% 2, 4, 6, 7. Combination chemotherapy with platinum agents, in spite of achieving higher response rates (about 30% in phase III trials), has not been shown to produce a survival benefit compared to single agents in randomized comparisons in recurrent/metastatic head and neck cancer 2, 4.

ELIGIBILITY:
Eligibility Criteria

Patients must have histologically or cytologically confirmed Squamous Cell Cancer of the Head and Neck either (a) metastatic (i.e. American Joint Committee on Cancer Staging System, 6th edition, stage IVC) or (b) recurrent, judged incurable by surgery or radiation.

Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with CT scan). RECIST criteria will be used (see section 9).

Therapeutic history in conformance with the following:

No more than one prior adjuvant/neoadjuvant chemotherapy and/or concomitant chemoradiotherapy regimen that may have included biologic/targeted agent.

No more than one prior regimen (chemotherapy or biologic/targeted) for recurrent/metastatic disease

ECOG performance status of 0-2 (Karnofsky > 60%; see Appendix A).

Patients must have normal organ and marrow function as defined below:

absolute neutrophil count > 1,000/L platelets > 75,000/L total bilirubin within normal institutional limits

AST(SGOT)/ALT(SGPT) 5 X institutional upper limit of normal creatinine within normal institutional limits

OR

creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

Urine protein should be screened by urine analysis for Urine Protein Creatinine (UPC) ratio (see Appendix). For UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be <1000 mg for patient enrollment.

Note: UPC ratio of spot urine is an estimation of the 24 urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is calculated using on of the following formula:

[urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/Dl [(urine protein) x0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L

All patients should have baseline tumor tissue available for EGFR determination (therapeutic target of cetuximab) and biomarker studies. Patients without available tissue at baseline may undergo tumor biopsy. Patients who provide consent and have accessible tumors will have a repeat biopsy 14 days (an interval between 12-16 days is acceptable) post initiation of therapy. Priority for study entry will be given to patients with easily accessible tumor and who consent to repeat biopsy. Study entry will not be restricted to patients who agree to further biopsies. If a patient enrolls on study and later refuses biopsy (excluding diagnostic), he/she may remain on study.

No prior treatment with cetuximab or bevacizumab or other EGFR or VEGF targeting agents.

Patients should not have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) and biologic/targeted agents within 3 weeks. At least 3 months should have elapsed after prior therapy with monoclonal antibodies.

At least 3 weeks should have elapsed from prior radiotherapy.

Patients must have no history of gross hemoptysis (defined as bright red blood of a ½ teaspoon or more) or coagulopathy. Patients with history of major tumor-related bleeding that is not controlled despite locoregional treatment or at high risk of recurrent tumor-related bleeding will be excluded.

Patients should not have a history of thrombosis (e.g. pulmonary embolism or deep venous thrombosis) and should not be on therapeutic anticoagulation (prophylactic use of warfarin 1 mg per day is allowed) and INR should be less than 1.5 at registration.

Patients with history of hypertension must be well-controlled (≤150/100) on a stable regimen of anti-hypertensive therapy.

Patients with tumors that invaded major vessels (e.g. the carotid) as shown unequivocally by imaging studies will be excluded due to the possibility of increased risk for tumor bleeding with bevacizumab therapy.

No major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or anticipation of need for major surgical procedure during the course of the study. No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to registration. No serious non-healing wound, ulcer, or bone fracture.

No unstable angina or myocardial infarction within the previous 6 months; no uncontrolled hypertension; no symptomatic congestive heart failure; no serious cardiac arrhythmia requiring medication; no clinically significant peripheral vascular disease; no history of any CNS cerebrovascular ischemia or stroke within the last 6 months; no active serious infection.

No other coexisting medical condition that would preclude full compliance with the study.

Patients may not be receiving any other investigational agents.

Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because of increased risks with bevacizumab.

Patients should not have a history of prior severe infusion reaction to a monoclonal antibody. Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies.

No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, unless there is a 3-year disease-free interval.

Age > 18 years. Because no dosing or adverse event data are currently available on the use of cetuximab and bevacizumab in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.

Ability to understand and the willingness to sign a written informed consent document.

Pregnant women are excluded from this study because cetuximab and bevacizumab have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cetuximab and bevacizumab, breastfeeding should be discontinued if the mother is treated with cetuximab and bevacizumab. The effects of cetuximab and bevacizumab on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately.

HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with cetuximab and bevacizumab. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

Inclusion of Women and Minorities

Both men and women and members of all ethnic groups are eligible for this trial. The proposed study population is illustrated in the table below.

Inclusion of Women in Plan: The gender distribution of our head and neck cancer patients is detailed in the table below. All efforts are made to recruit women patients with head and neck cancer to the University of Pittsburgh Medical Center.

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gibson, MD, Principal Investigator — Eastern Cooperative Oncology Group
Locations (4):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - Case Western Reserve University, Cleveland, Ohio
  - UPMC / UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson, Houston, Texas

REFERENCES:
- [Result] Argiris A, Kotsakis AP, Hoang T, Worden FP, Savvides P, Gibson MK, Gyanchandani R, Blumenschein GR Jr, Chen HX, Grandis JR, Harari PM, Kies MS, Kim S. Cetuximab and bevacizumab: preclinical data and phase II trial in recurrent or metastatic squamous cell carcinoma of the head and neck. Ann Oncol. 2013 Jan;24(1):220-5. doi: 10.1093/annonc/mds245. Epub 2012 Aug 16. PMID 22898037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We report results in 46 eligible patients. Two patients were deemed ineligible, one because subsequent biopsy showed that measurable disease was actually steoradionecrosis and not recurrent laryngeal cancer. The other patient required surgery for cholecystitis before starting treatment; this patient never initiated protocol treatment.
Groups:
- Cetuximab Plus Bevacizumab: Cetuximab plus bevacizumab
  Cetuximab: • Cetuximab 400 mg/m2 IV over 120 minutes on day 1 of cycle 1 ONLY
  • Cetuximab dose will be 250 mg/m2 IV over 60 minutes weekly on ALL subsequent administrations
  Bevacizumab: Once every 3 weeks, 15 mg/kg of bevacizumab will be given by IV infusion after cetuximab has been given
Period: Overall Study
Arm/Group | Cetuximab Plus Bevacizumab
Started | 46
Overall Response Rate | 7
Completed | 45
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: STARTED 46; Overall Response Rate 7; COMPLETED 45; Not Completed 1
Arm/Group | Cetuximab Plus Bevacizumab
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: Years] | 61.5 [33 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46
Primary disease site [Number; unit: participants]
  Oropharynx | 17
  Oral cavity | 14
  Larynx | 7
  Others | 8
Recurrent disease [Number; unit: participants] | 44
Prior radiation [Number; unit: participants] | 44
Prior surgery [Number; unit: participants] | 30
Prior chemotherapy [Number; unit: participants]
  Prior chemotherapy | 42
  1 prior palliative regimen | 17
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) criteria: 0-Fully active. 1-Ambulatory, carry out work of a light or sedentary nature. 2=Ambulatory, capable of all self care. 3-Capable of limited self care, confined to bed or chair more than 50% of waking hours. 4-Completely disabled, no self care, totally confined to bed or chair. 5-Dead.
  participants
    0 | 11
    1 | 31
    2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is the percentage of patients whose cancer shrunk or disappeared after study treatment. ORR was determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) : Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Progressive Disease (PD): at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 5 years
Population: Assess all patients included in this study for response to treatment, per protocol. Of 46 eligible patients, 45 were evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Bevacizumab
Number analyzed (Participants) | 45
percentage of participants | 16 [7 to 24]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is the length of time during and after treatment that patients are alive with the disease but it does not get worse. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI), Progressive Disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Up to 5 years
Population: All patients included in study are assessed for response to treatment, per protocol. Of 46 eligible patients, 45 were evaluable for response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab Plus Bevacizumab
Number analyzed (Participants) | 45
Months | 2.8 [2.7 to 4.2]

3. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of study/treatment that diagnosed patients are still alive.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Bevacizumab
Number analyzed (Participants) | 45
months | 7.5 [5.7 to 9.6]

4. Secondary Outcome: Change in Serum Cytokine Concentrations
Description: Ratio of serum cytokines concentration after treatment with cetuximab and bevacizumab to baseline serum cytokines concentration, in picogram/milliliter (pg/ml) for 13 different cytokines. [post-treatment (pg/ml) / baseline (pg/ml)]
Time Frame: Up to 5 years
Population: Patients treated with cetuximab and bevacizumab who provided baseline and post-treatment serum samples.
Measure: Number; unit: post-treatment/baseline pg/ml ratio
Arm/Group | Cetuximab Plus Bevacizumab
Number analyzed (Participants) | 20
post-treatment/baseline pg/ml ratio
  TGFa | 3.3711
  PIGF | 1.9453
  VEGF | 0.1203
  EGFR | 1.5875
  IP.10 | 1.25
  VEGFR.2 | 1.1032
  FGFb | 0.7346
  FGFa | 0.0000
  IL.6 | 1.3831
  HGF | 0.9622
  GCSF | 1.2652
  EGF | 0.7878

5. Secondary Outcome: Disease Control Rate (DCR) ((Clinical Benefit Rate (CBR))
Description: Disease Control Rate (DCR) (or Clinical Benefit Rate (CBR)), is defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to cetuximab and bevacizumab.
  DCR = number of patients with (at least) partial response or stable disease / total number of evaluable patients
Time Frame: At 12 weeks
Population: Patients that were evaluable for 'best response' to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cetuximab Plus Bevacizumab
Number analyzed (Participants) | 45
percentage of participants | 73

ADVERSE EVENTS:
Arm/Group | Cetuximab Plus Bevacizumab
Serious Adverse Events (participants affected / at risk) | 22/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Bevacizumab (N=46)
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 7
Stricture/stenosis (including anastomotic), GI, Esophagus (Gastrointestinal disorders) | 1
Stricture/stenosis (including anastomotic), GI, Pharynx (Gastrointestinal disorders) | 1
Pain, Abdomen NOS (Gastrointestinal disorders) | 2
Hemorrhage, pulmonary/upper respiratory, Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Infection with Grade 3 or 4 neutrophils, Lung (pneumonia) (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Infection with unknown ANC, Esophagus (Infections and infestations) | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Mood alteration, Depression (Psychiatric disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Pain, Head/headache (Nervous system disorders) | 1
Pain, Oral cavity (Gastrointestinal disorders) | 1
Pain, Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Pain, Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction/stenosis of airway, Larynx (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Bevacizumab (N=46)
Anemia (Blood and lymphatic system disorders) | 11
Cardiac disorders - Other (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
External ear pain (Ear and labyrinth disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 2
Cataract (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 2
Eye disorders - Other (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eyelid function disorder (Eye disorders) | 2
Watering eyes (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 17
Esophageal pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 22
Oral hemorrhage (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 14
Rectal hemorrhage (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Chills (General disorders) | 7
Edema face (General disorders) | 6
Edema limbs (General disorders) | 2
Facial pain (General disorders) | 2
Fatigue (General disorders) | 31
Fever (General disorders) | 7
General disorders and administration site conditions - Other (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 10
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 2
Bronchial infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Esophageal infection (Infections and infestations) | 1
Gum infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 5
Joint infection (Infections and infestations) | 1
Lip infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 2
Nail infection (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Skin infection (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Injury to jugular vein (Injury, poisoning and procedural complications) | 1
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1
Intraoperative head and neck injury (Injury, poisoning and procedural complications) | 1
Venous injury (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 5
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 11
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Trismus (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 4
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 20
Nervous system disorders - Other (Nervous system disorders) | 3
Neuralgia (Nervous system disorders) | 1
Olfactory nerve disorder (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Trigeminal nerve disorder (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 7
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 7
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 19
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Nail loss (Skin and subcutaneous tissue disorders) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 12
Rash acneiform (Skin and subcutaneous tissue disorders) | 32
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 8
Skin ulceration (Skin and subcutaneous tissue disorders) | 5
Flushing (Vascular disorders) | 2
Hematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 3
Peripheral ischemia (Vascular disorders) | 1
Vascular disorders - Other (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less